CLINICAL TRIAL: NCT00085761
Title: An International, Multicenter, Randomized, Double-Blind, 12-Week Controlled Study of NGX-4010 for Treatment of Painful HIV-Associated Neuropathy
Brief Title: Study of NGX-4010 for Treatment of Painful HIV-Associated Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated in view of the C107 findings demonstrating efficacy at doses of 90 and 30 minutes
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C112
Record Dates: First submitted 2004-06-14; First posted 2004-06-17 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections; Peripheral Nervous System Diseases; Pain
Keywords: Dermal assessment; Pain measurement; Diary; Neuropathy; Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; HIV Infections/*complications/*drug therapy; Pain; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Pain

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is to determine if an investigational drug, NGX-4010 (high-concentration capsaicin patch), is safe, tolerable and effective in treating painful HIV-associated neuropathy.

ELIGIBILITY:
Key Eligibility Criteria:

* Must have had HIV-associated neuropathy for at least 2 months, with moderate to severe pain in both feet.
* Must not have significant pain in feet due to other causes (for example, arthritis).
* Must have intact skin at the treatment area.
* Must be prepared to remain on the same pain medications at the same doses as before the study for the entire duration of the study (12 weeks).
* Must not use topical pain medications for HIV-associated neuropathy.
* Must be able to comply with study requirements such as completing daily pain diary and attending study visits.
* Must be at least 18 years old, not pregnant, and be able to take care of self independently, with only occasional assistance if needed.
* No significant medical problems of the heart, kidneys, liver or lungs, or cancer.
* No history or current problem with substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NeurogesX Investigational Site, Sarasota, Florida
  - NeurogesX Investigational Site, Annandale, Virginia